CLINICAL TRIAL: NCT03092661
Title: Reference Data for Neonatal Oxygen Saturation - a Pilot Study.
Brief Title: Baby Oxygen Saturation Study
Acronym: BOSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: GN16RM676P
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Normative Oxygen Saturation Levels in Infants
Keywords: Oxygen saturation; Pulse oximetry; Neonate; Infant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To define preliminary reference (normative) limits for healthy, newborn baby oxygen saturation parameters using the Masimo Radical 7® monitor.

To assess protocol feasibility in terms of acceptability to parents and infants.

To inform the design of a future larger study where reference limits will be fully defined across a wider gestational age group.

DETAILED DESCRIPTION:
Blood oxygen saturation is the percentage of haemoglobin carrying oxygen. It is accepted that healthy term infants breathing room air have oxygen saturation levels of 95% or greater, similar to adults (Levesque 2000). Blood oxygen saturation levels have to be carefully balanced in infants who are born prematurely. High saturation levels are associated with retinopathy of prematurity (ROP) and lower saturation levels with increased mortality (SUPPORT 2010; BOOST II 2013).

Current practice is to maintain premature infants' oxygen saturations between 88 and 93%. After 36 weeks' postmenstrual age, the risk of ROP is greatly reduced and these target oxygen saturations are typically increased to greater than 93%. Lower saturations beyond this time are associated with poor weight gain and are considered to carry a risk of developing pulmonary hypertension (Poets 1998). Many of the smallest and most premature infants will continue to require supplemental inspired oxygen after 36 weeks' postmenstrual age in order to maintain saturations greater than 93%, so called "chronic lung disease of prematurity". Some of these infants will require to be discharged home on supplemental oxygen. The need for home oxygen is determined by measurement of pulse oximetry prior to discharge.

A recently developed device, the Masimo Radical 7, is now in widespread use in preterm infants nearing discharge from the neonatal unit. This device is more accurate (Bohnhorst 2002), derives extra physiological measures from the oxygen saturation data (heart rate and perfusion index) and offers longer-term data storage than other models currently in clinical use. In addition, the Masimo Radical 7 with its analysis software is capable of counting and measuring shorter-term dips in oxygen saturation (Sedowofia 2008). An oxygen saturation study can be measured in terms of the overall oxygen saturation, and/or the number, duration and severity of these dips. Increasing use of the Masimo Radical 7 to record oxygen saturation studies in preterm infants nearing discharge from the neonatal unit has, for a significant number of infants, revealed more than previously suspected episodes of reduced oxygen saturation which are frequently not clinically apparent. Because of a dearth of data recorded from healthy term babies in the immediate newborn period, the "normal" Masimo Radical 7 trace is not well defined and the significance of these short dips in oxygen saturation is not clear. Defining acceptable saturation limits depends on a complete understanding of what is normal: in other words, deriving adequate reference limits from hundreds of healthy neonates (CLSI 2008; Pan 1990).

Multiple studies of oxygen saturation levels in neonates have been conducted, but disparate devices and protocols, and heterogeneity in age, gestation and morbidity of subjects preclude any universal clinical decision limit for normal oxygen saturation profile in prematurely-born neonates. Furthermore, as noted above, most currently-used oxygen saturation monitors do not capture very short-term changes in oxygen saturation.

This study will define preliminary reference limits for pulse oximetry in newly born healthy term babies, in order better to be able to interpret oxygen saturation recordings made in preterm babies nearing term corrected age and hospital discharge. The investigators will assess feasibility of data collection, and use the data to inform a subsequent larger study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term baby admitted to postnatal ward of Princess Royal Maternity.
* Written informed parental consent.
* Delivery by elective caesarean section.

Exclusion Criteria:

* Significant congenital abnormality.
* Any respiratory or cardiac concerns.
* Treatment for suspected sepsis.

Ages: 1 Hour to 1 Month | Sex: All
Age Groups: Child
Study Population: The study will complete oximetry measurements from 40 newborn infants, recruited at the Princess Royal Maternity.
  Study participants will be newly born, healthy, appropriately grown, term infants delivered by elective caesarean section. These infants will generally be around 39 weeks' gestation.
  This group has been chosen due to their tightly grouped gestational and postnatal age ranges with the aim of reducing variability related to age or maturity. Pragmatically, mothers undergoing delivery by caesarean section are likely to remain in the hospital for 38-45 hours, thus participation in an oximetry study will not delay discharge.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-03-27 (Actual); Primary Completion 2018-01-31 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
Oxygen saturation graph | up to 24 hours
  A trend graph of saturation and heart rate for the recording.
Oxygen saturation summary statistics. | up to 24 hours
  Statistics describing the distribution of the saturation trend recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Mactier, MD, Principal Investigator — Helen.Mactier@ggc.scot.nhs.uk
Locations (1):
- Princess Royal maternity, Glasgow, Scotland, United Kingdom